CLINICAL TRIAL: NCT05738538
Title: Expanded Access to Ziftomenib
Status: Available | Type: Expanded Access
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Expanded Access to Ziftomenib
Record Dates: First submitted 2023-02-10; First posted 2023-02-22 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia, With Appropriate Mutations; Acute Myeloid Leukemia, With NPM1 Mutations
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ziftomenib

SUMMARY:
Requests for single patient expanded access to ziftomenib monotherapy may be considered for eligible adult patients with Acute Lymphoblastic Leukemia (ALL) with KMT2A rearrangements, or Acute Myeloid Leukemia (AML), with NPM1 mutations or KMT2A rearrangements.

To request access, use Responsible Party contact information provided in this record.

Expanded access for ziftomenib is only available in the United States.

DETAILED DESCRIPTION:
• Subsection Condition:

* NPM1 mutation in AML patients
* KMT2A rearrangement in AML patients
* KMT2A rearrangement in ALL patients

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Diagnosed with Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL).
* Adult, ages 18+.
* Has exhausted appropriate standard treatments without success and no comparable or satisfactory alternative treatment is available or exists to treat the disease or condition. For newly diagnosed AML patients with either NPM1-mutant, or KMT2A-rearranged AML, ziftomenib therapy will be considered for patients not eligible for ongoing clinical trials. In the case of patients with KMT2A-rearranged AML, Expanded Access to ziftomenib will only be provided for use in combination with FDA-approved therapies currently under clinical investigation at Kura Oncology (e.g., venetoclax + azacitidine, cytarabine + daunorubicin).
* Is ineligible for participation in any ongoing clinical study of the investigational drug, which includes lack of access due to geographic limitations.
* Meets any other pertinent medical criteria for access to the investigational drug, as established by Kura Oncology.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult